CLINICAL TRIAL: NCT05400551
Title: Epidemiology of Craneofacial Injuries in Rink Hockey Athletes
Brief Title: Craneofacial Injuries in Rink Hockey Athletes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Principal Investigator, University of Oviedo
Other Study IDs: UO2022-01
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Head Injury; Face; Concussion, Brain
Keywords: rink hockey; injury; epidemiology; burden
MeSH Terms: conditions — Craniocerebral Trauma; Facies; Brain Concussion; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To collect the number of injuries that affect the face and head in rink hockey athletes prospectively during a regular season.

DETAILED DESCRIPTION:
To collect the number of injuries that affect the face and head in rink hockey athletes prospectively during a regular season, while collecting athlete´s exposure and specifical injury characteristics (Burden, mechanism, situation, etc)

ELIGIBILITY:
Inclusion Criteria:

* Compete in a spanish rink hockey league
* play at least in one game during ther regular season

Exclusion Criteria:

* do not accept the participation in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: athletes that compete in rink hockey, independently of their age or sex
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants injured | september 2022 to march 2023
  nº of injuries affecting the head or face per time (X/1000h)
days lost due to injury | september 2022 to march 2023
  nº of days lost due to injury affecting the head or face per time (X days/1000h)

SECONDARY OUTCOMES:
usage of helmet | september 2022 to march 2023
  characterise if the player was using a helmet or not when the injury happened
situational characteristics of the injury | september 2022 to march 2023
  register when the injury happened (training or game)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hugo Olmedillas, Oviedo, Principality of Asturias
  - Universidad de Oviedo, Oviedo, Principality of Asturias

IPD SHARING:
Plan to Share IPD: Undecided